CLINICAL TRIAL: NCT03087734
Title: Evaluation of a New Model of Metallic Bar and Stabilizer for Use in the Minimally Invasive Repair of Pectus Excavatum
Brief Title: Evaluation of a New Model of Metallic Bar and Stabilizer for Use in MIRPE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Principal Investigator, Miguel L. Tedde, Principal Investigator, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2014/15290-7
Record Dates: First submitted 2016-10-24; First posted 2017-03-22 (Actual); Last update posted 2021-10-12 (Actual); Status verified 2021-10

CONDITIONS: Funnel Chest
Keywords: Prostheses and Implants
MeSH Terms: conditions — Funnel Chest

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Perpendicular stabilizer (Active Comparator): Implantation of regular bar with perpendicular stabilizers
  Interventions: Device: Implantation of regular bar with perpendicular stabilizers
- Oblique stabilizer (Experimental): Implantation of new model of bar with oblique stabilizers
  Interventions: Device: Implantation of new model of bar with oblique stabilizers

INTERVENTIONS:
Device: Implantation of new model of bar with oblique stabilizers — Implantation of new model of bar with oblique stabilizers
  Arms: Oblique stabilizer
Device: Implantation of regular bar with perpendicular stabilizers — Implantation of regular bar with perpendicular stabilizers
  Arms: Perpendicular stabilizer

SUMMARY:
Pectus excavatum (PE) is the most common deformity of the chest wall, occurring in approximately 1/1000 people. Currently, surgical treatment by minimally invasive technique is consolidating as preferred technique for the treatment of this condition. In this technique a metal bar is inserted in retrosternal position, pushing the sternum without the necessity of resecting the condral cartilages. Despite the advantages obtained with this technique, it is not without complications and the displacement of the bar is one of the most important. In order to minimize this problem we developed a new model of stabilizers, as well as all necessary instruments for performing minimally invasive surgery. The aim of this study is to compare two surgical groups, one making use of the new oblique stabilizer compared to the conventional perpendicular stabilizer to determine which one has less displacement. Furthermore, this study also aims to assess the full range of instruments developed by a national company, to carry out this type of surgery, which has cost compatible with our economic reality, and that can be accessible to our Public Health patients.

DETAILED DESCRIPTION:
Introduction Pectus excavatum (PE) is presented as a sunken sternum in the midline and these chest deformities are not uncommon, occurring in approximately 1/1000.

It is commonly accepted that the abnormal growth of condral cartilage results in displacement of the sternum. Most patients and their parents seek medical advice for psychosocial concerns, particularly related to the cosmetic aspects and the consequent aversion to sports or public exposure. Physiological tests are often normal, but both the cardiac index and pulmonary function may be affected.

Surgical treatment of pectus excavatum Nuss broke the paradigm in PE surgery with the publication of their results using a technique called minimally invasive. This technique involves lateral incisions in the chest and the placement of one or two temporary steel bars, which are shaped during surgery, specifically for each patient. These bars are placed in retrosternal position and the sternum is elevated without the need of cartilage resection.

This surgical technique, in addition to the bars and stabilizers, needs a set of instruments that are used in the customization of the bar for each patient and, after three years, the withdrawal of the bar at the end of the treatment.

Another problem refers to the displacement of the metallic bars that are positioned under the sternum and that are held in position by placing stabilizers, one at each lateral end of the bar. These stabilizers, which are perpendicular to the bar, has the function to expand its area of contact with the chest wall in order to prevent it from moving from its position.

In order to increase the stability of the bar, preventing their movement, various modifications have been proposed. The investigators believe that further modification can be introduced. If the stabilizer metal bar has an oblique position relative to the bar (rather than perpendicular as it is currently) it will be perpendicular to the ribs, thus increasing its area of contact with the chest wall, which might bring more stability.

The investigators are also proposing that the new metal bar that is being developed is completely smooth, not having the usual slots that the current model has at the extremities of the bars. The reason for this is to try to prevent bleeding during bars withdrawal after 3 years of use.

Another proposed amendment is a pressure screw incorporated into the stabilizer itself.

Search object The object of research is the development of a new model of metallic bar and stabilizers, as well as dedicated surgical instruments whose purpose is to perform minimally invasive repairs of PE.

Social relevance One of the reasons why the Public Health in Brazil gives no coverage for this type of surgical treatment for patients with PE is the high cost of surgical equipment that is imported. The development of this material in the country, as is being proposed in this project, has high social relevance that may represent savings by avoiding the purchase of imported material and the possibility of making available this type of surgical treatment for patients served by our public health.

Site of the search The research will be performed in the Department of Thoracic Surgery, Heart Institute (InCor) of the Hospital das Clinicas, Faculty of Medicine, University of São Paulo.

ELIGIBILITY:
Inclusion Criteria:

* Pectus excavatum patients

Exclusion Criteria:

* Presence of complex congenital anomalies;
* Retardation neurodevelopment;
* Congenital heart disease;
* Chronic Immunosuppression.

Min Age: 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-10-03 (Actual); Primary Completion 2018-09-25 (Actual); Study Completion 2019-03-01 (Actual)

PRIMARY OUTCOMES:
Grade of metallic bar dislodgment measured through Rx images | One year
  The grade of metallic bar dislodgment will be measured through the comparison of the Rx taken in patient follow up in terms of: a) bar flipping; b) lateral sliding and c) hinge-point disruption

CONTACTS AND LOCATIONS:
Overall Officials: Paulo M Pego-Fernandes, Study Chair — Heart Institute (InCor), Hospital das Clinicas, University of Sao Paulo
Locations (1):
- Heart Institute (InCor) Hospital das Clinicas da Faculdade de Medicina da Universidade de Sao Paulo, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tedde ML, De Carvalho RLC, De Campos JRM, Da Silva DAG, Okumura EM, Guilherme GF, Marchesi AC, Petrizzo P, Souto Maior BS, Pego-Fernandes PM. Randomized comparison of oblique and perpendicular stabilizers for minimally invasive repair of pectus excavatum. Interdiscip Cardiovasc Thorac Surg. 2024 Mar 5;38(3):ivae040. doi: 10.1093/icvts/ivae040. PMID 38492558